CLINICAL TRIAL: NCT06397846
Title: Identification of Biomarkers Associated With the Presence of Malignant Pancreatic Lesions Compared to Benign Lesions.
Acronym: PANORAMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023/842
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Benign Pancreatic Lesion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological sample (Experimental): Blood sample
  Interventions: Other: Biological sample

INTERVENTIONS:
Other: Biological sample — blood sample will be collected at baseline

SUMMARY:
The challenge for medical oncology is to develop plasma biomarkers that can detect the influence of the stroma on diagnosis, prognosis and response to chemotherapy.

Today, there is no validated blood test to help diagnose pancreatic cancer (PDAC). The search for blood biomarkers of the tumor stroma and immunological markers is therefore a major challenge in orienting the diagnosis towards PDAC and optimizing the therapeutic management of pancreatic cancers.

The aim of the study is to identify biomarkers associated with the presence of malignant pancreatic lesions (patients from the Pancreas-CGE cohort, a cohort already set up by our team) compared with benign lesions (patients followed up for benign pancreatic lesions). Candidate biomarkers from our preliminary work will be considered initially. Other biomarkers may be explored secondarily.

The ultimate goal is to develop a clinico-biological signature that is as efficient as possible in predicting the presence of malignant pancreatic lesions compared with benign ones.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥18 years
* Patient followed for benign pancreatic lesions:

chronic pancreatitis acute pancreatitis at a distance from the acute episode (> 4 weeks) with indication for echo-endoscopy for suspected precancerous pancreatic lesions (PanIN, TIPMP, mucinous cystadenomas) or other cystic lesions (serous cystadenomas)

Exclusion Criteria:

* Malignant pancreatic tumor
* Legal incapacity or limited legal capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
the malignant versus benign nature of the pancreatic lesion, based on radiological, echo-endoscopic and/or anatomopathological characteristics. | one visit at baseline

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - University Hospital of Besancon, Besançon
  - Hôpital Nord Franche-Comté, Montbéliard